CLINICAL TRIAL: NCT02107547
Title: Evaluation of Biceps Tenodesis vs Labral Repair for Type 2 Superior Labrum Anterior and Posterior Lesions, A Randomized Controlled Trial
Brief Title: Outcomes of Biceps Tenodesis or Labral Repair for Treatment of Type 2 Superior Labrum Anterior and Posterior Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 13-0085
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Type 2 SLAP Lesions
Keywords: Randomized Controlled Trial (RCT); Type 2 SLAP lesions; labral tear; biceps tenodesis; shoulder surgery; RCT; Comparison between two alternative surgical procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biceps tenodesis (Active Comparator): 32 subjects in the study will receive biceps tenodesis as a surgical intervention
  Interventions: Procedure: Biceps tenodesis
- Labral repair (Active Comparator): 32 subjects in the study will receive labral repair as a surgical intervention
  Interventions: Procedure: Labral repair

INTERVENTIONS:
Procedure: Biceps tenodesis — A biceps tenodesis involves cutting the tendon within the shoulder joint and reattached further down the arm.
  Arms: Biceps tenodesis
Procedure: Labral repair — Repair of a Superior Labrum Anterior and Posterior lesion involves placing small anchors in the glenoid to re-attach the torn labrum.
  Arms: Labral repair

SUMMARY:
The purpose of the study is to determine which of the two alternative surgical interventions (biceps tenodesis or labrum repair surgery) is better in the treatment of Type 2 Superior Labrum Anterior and Posterior lesions.

DETAILED DESCRIPTION:
The labrum is a structure which provides stability to the shoulder joint. A superior labral tear from anterior to posterior lesion is an injury to the labrum at the insertion of the biceps muscle. The grading system is related to the severity of the tear. A type 2 tear is an intermediate grade tear. These are commonly treated in two ways: either by repairing the labrum with bone anchors or by cutting the biceps tendon and re-affixing it more distally. No method has been shown to be superior to the other and surgeons generally choose to proceed however they are most comfortable. The study will seek to determine how these injuries are best treated. Inclusion criteria: patients with type 2 superior labral tear from anterior to posterior tears who are under the age of 45. Throwing athletes are excluded due to their unique demands.

Subjects will be randomly assigned to one of two groups. Prior to surgery patients will be evaluated in clinic, full histories and physicals will be performed and their functional status will be evaluated using validated questionnaires including the American Shoulder and Elbow Society score and quality of life measurements.

Both groups will be treated first with a shoulder arthroscopy. The experimental portion of the study will involve whether the patient is then treated with repair of the Superior Labrum Anterior and Posterior lesion or with tenodesis. Repair of a Superior Labrum Anterior and Posterior lesion involves placing small anchors in the glenoid to re-attach the torn labrum. A biceps tenodesis involves cutting the tendon within the shoulder joint and reattached further down the arm. Physical therapy will be initiated after surgery and will be identical in both groups. It will be recommended but not required as part of the study. Progress notes, operative reports, and questionnaires will also be retained as part of the study. Patients will be in a sling for the first 4 weeks after surgery. Post-operatively, physical examinations findings and American Shoulder and Elbow Surgeons scores at 3, 6, and 12 months. These will be compared to the preoperative results and to the other experimental arm of the study. Post-operative imaging will not be obtained. No computerized tomographies will be required as part of the study. No Magnetic Resonance Imagings will be required as part of the study--patients enrolled in the study will likely have had an MRI performed outside of the study period to determine if they have an isolated Superior Labrum Anterior and Posterior tear but no MRIs will be performed as part of the study. No lab reports or Physical therapy reports will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with MRI diagnosed Superior Labrum Anterior and Posterior 2 lesion

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | one year
  The scale measures pain from 0 to 10 and also includes a questionnaire for assessing the activity of daily living.

SECONDARY OUTCOMES:
EuroQol five dimensions | one year
  The questionnaire measures mobility, ability to care for self, ability to perform usual activities, pain/discomfort, and anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Lewis L Shi, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No